CLINICAL TRIAL: NCT04810572
Title: Evaluation of the Effects of a Nutraceutical Composition Containing Derivatives From Natural Products on the Modulation of the Endocrine Neuroimmune Axis - Translational Study.
Brief Title: Nutraceutical Composition Containing Natural Products Derivatives on the Modulation of the Endocrine Neuroimmune Axis
Acronym: NCCNPDMENA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ana Flávia Marçal Pessoa, Principal Investigator, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 39984320.5.0000.0068
Record Dates: First submitted 2021-02-20; First posted 2021-03-23 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Insulin Resistance; Inflammatory Bowel Diseases; Overweight and Obesity; Healthy
MeSH Terms: conditions — Insulin Resistance; Inflammatory Bowel Diseases; Overweight; Obesity | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 - composition with Silymarin (L5-Plus) (Active Comparator): This group compound with healthy and overweight/obese-I will receive the composition with Silymarin (Silybum marianum), in a diary dose of 140 mg for 180 days.
  The formulation of the supplement/composition (Patent number: BR 10 2020 016156 3).
  Interventions: Dietary Supplement: Composition with Silymarin; Dietary Supplement: Low-mineral composition without Silymarin
- Group 2 - composition without Silymarin (L5-Plus) (Active Comparator): This group compound with healthy and overweight/obese-I will receive the composition without Silymarin (Silybum marianum), in a diary dose for 180 days.
  The formulation of the supplement/composition (Patent number: BR 10 2020 016156 3).
  Interventions: Dietary Supplement: Composition with Silymarin; Dietary Supplement: Low-mineral composition without Silymarin
- Group3 - Low-mineral composition without Silymarin (L5) (Active Comparator): This group compound with healthy and overweight/obese-I will receive the composition without Silymarin (Silybum marianum), in a diary dose for 180 days.
  The formulation of the supplement/composition (Patent number: BR 10 2020 016156 3).
  Interventions: Dietary Supplement: Composition with Silymarin; Dietary Supplement: Low-mineral composition without Silymarin

INTERVENTIONS:
Dietary Supplement: Composition with Silymarin — Volunteers will receive supplementation for 180 days. They took 4 capsules daily. Two capsules in the morning and two capsules at night.
  There will be blood and feces collection at zero time, before supplementation, after 30, 90 and 180 days from the beginning of supplementation.
  Other Names: Patent number: BR 10 2020 016156 3
Dietary Supplement: Low-mineral composition without Silymarin — Volunteers will receive supplementation for 180 days. They took 4 capsules daily. Two capsules in the morning and two capsules at night.
  There will be blood and feces collection at zero time, before supplementation, after 30, 90 and 180 days from the beginning of supplementation.

SUMMARY:
The use of natural products in the prevention or treatment of chronic diseases is an emerging field in current medicine. And studying the mechanisms of actions by which natural products act in our bodies contributes to the rational use of these products. And the combination of different natural products such as prebiotics (FOS- fructooligosaccharides, GOS-Galactooligosaccharides and beta-glucans derived from yeast), herbal medicine (Silybum marianum), and minerals (Se-selenium, Zn-Zinc, and Mg-Magnesium), o which would result in a synergistic association between them can contribute to achieving not only preventive effects but treatment for chronic diseases such as diabetes and obesity. The present study aims to study the effects of a composition containing natural products on factors and markers that are part of mitochondrial biogenesis and the neuroimmune-endocrine system in healthy volunteers and that present grade 1 overweight/obesity.

DETAILED DESCRIPTION:
Obesity and diabetes are chronic diseases characterized by increased visceral adipose tissue and sub-acute inflammation. These conditions can lead to insulin resistance, hyperglycemia, oxidative stress], and lipotoxicity, and lead to the development of metabolic syndrome. Previous work has shown that these comorbidities, as well as high levels of glucocorticoids, can modulate the hypothalamic-pituitary-adrenal (HPA) axis and inflammatory response. In some cases, these conditions and responses perturb neuroimmune endocrine system homeostasis.

Another potential outcome arising from inflammation, insulin resistance, hyperglycemia, and lipotoxicity is a nonalcoholic fatty liver disease (NAFLD), a chronic liver disease that often coexists with obesity-related type 2 diabetes. Previous studies have demonstrated that NAFLD compromises glycemic and lipid homeostasis. The hyperglycemia and the lipotoxicity drive the metabolic pathways of the cell towards gluconeogenesis, glycolysis, and de novo lipogenesis, and the subsequent increase in free fatty acid (FFA) production can cause oxidative stress.

Previous studies have shown that non-pharmacological interventions can be used as strategies for treating and/or preventing inflammatory and metabolic diseases. Furthermore, exploiting specific proteins and transcription factors that target the mitochondria represents potential mechanisms for these interventions.

Along these lines, natural products and derivatives thereof, often referred to as natural medicines, have been gaining notoriety as sources of effective therapeutics. For example, polyphenols present in plants can be metabolized to form propionic acid, which is later transformed into another metabolite, butyrate. As reviewed by Juárez-Hernández et al., Na-butyrate and synthetic derivatives thereof increase prebiotic lactobacilli and bifidobacteria growth in the colon, consequently improving thermogenesis and energy expenditure, ultimately reducing hepatic lipid deposition, improving triacylglycerol content and insulin resistance and protecting against metabolic impairment, as well as liver inflammation and/or damage. Furthermore, butyrate can induce the expression of fibroblast growth factor 21 (FGF-21), which plays a vital role in stimulating hepatic fatty acid β-oxidation. In this sense, prebiotics may be a promising treatment for chronic inflammatory and metabolic diseases in humans.

The efficacy of prebiotic compounds, such as fructooligosaccharides (FOS), galacto-oligosaccharides (GOS) and yeast β-glucans, minerals including magnesium, zinc, selenium, and plants like Silybum marianum (L.) Gaerth. (Silymarin), have been evaluated for the treatment of specific diseases. However, most of these studies only describe the effects of the supplements being administered alone. Thus, the present study monitored the synergic effects of a novel supplement formulation containing prebiotics, yeast β-glucans, minerals, and silymarin on lipid metabolism, inflammatory and mitochondrial proteins in eutrophic, and overweight/obesity I volunteer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (healthy) and sedentary volunteers: people without chronic use of drugs for chronic inflammatory diseases that require the use of corticosteroids or NSAIDs (Non-Steroidal Anti-inflammatories) for a period of more than 15 days. BMI (Body Mass Index) of 24.9 Kg / m2.
* Sedentary overweight/obesity grade 1 volunteer: overweight people, with a BMI of 25.0 to 29.9 kg / m2; and grade 1 obesity with a BMI of 30.0 and 34.9 kg / m2, with or without dyslipidemia and/or non-insulin-dependent type 2 diabetics.

Exclusion Criteria:

* Volunteers who are allergic to some of the components of the nutraceutical formulation, who use insulin, corticosteroids, and NSAIDs for more than 15 days, AIDS, hepatitis, patients undergoing chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Change Lipid Profile Baseline after 4, 12 and 24 weeks of intervention. | Baseline and 4, 12 and 24 weeks.
  The serum levels of cholesterol (mg/dL), triglycerides (mg/dL), and high-density lipoprotein cholesterol (HDL-c) (mg/dL) will be measured with a commercially available kit (Bioclin, Belo Horizonte, MG, Brazil).
Change Lymphocyte Phenotype at 4, 12 and 24 weeks after intervention. | Baseline and 4, 12 and 24 weeks.
  Lymphocytes will be isolated from 12 mL of whole blood. Anticoagulated blood is layered onto Histopaque-1077. During centrifugation, erythrocytes are aggregated by polysucrose and rapidly sediment. Lymphocytes and other mononuclear cells remain at the plasma/ Histopaque-1077 interface.
  Single-cell suspensions with lymphocyte will be incubated with the human antibodies indicated:
  * T helper type 1 (Th1) cells are a subset of CD4+ effector T cells (cell surface expression of IL-12 R beta 2, IL-27 R alpha/WSX-1, IFN-gamma R2, IL-18 R, CCR5, and CXCR3);
  * T helper type 2 (Th2) cells are a subset of CD4+ effector T cells (cell surface markers CCR3, CCR4, CCR8, CXCR4, and ST2/IL-1 R4).
  * T helper type 9 (Th9) cells are a subset of CD4+ effector T cells [helper cell subsets including T-bet (Th1 cells), GATA-3 (Th2 cells), ROR gamma t (Th17 cells), or FoxP3 (regulatory T cells)].
  Cells will be analyzed in a FACSCalibur (BD Biosciences, San Diego, CA).
Change Serum Cortisol Level Baseline after 4, 12 and 24 weeks of intervention. | Baseline and 4, 12 and 24 weeks.
  Serum cortisol (pg/ml) will be measured by Elisa Kit (Cayman Chemical, Ann Arbor, MI, USA), according to the recommendations of the manufacturer.
Change Gut Microbiota Baseline after 4, 12 and 24 weeks of intervention. | Baseline and 4, 12 and 24 weeks.
  For analysis of the gut microbiota, stool samples will be collected (approximately 15g) in a sterile plastic tube kit (ColOff®) and kept frozen at -80°C until the DNA extraction procedure. The material will not be collected in cases of watery stools or when the evacuation was not spontaneous (use of laxatives for evacuation). At the time of stool collection, none of the participants should be using or has used antibiotics for at least one month. Samples will be collected before bowel preparation for surgery, if necessary. Genomic DNA will be extracted from the fecal contents using the QIAamp DNA Stool Mini Kit (Qiagen, Hilden, Germany) according to the manufacturer's instructions and the microbiota composition analysis will be performed by 16S rRNA gene sequencing on the Illumina MiSeq platform.
Change Haemogram Parameters Baseline after 4, 12 and 24 weeks of intervention. | Baseline and 4, 12 and 24 weeks.
  Anticoagulated blood will be used to do the complete blood count performed using basic laboratory equipment or an automated hematology analyzer, which counts cells and collects information on their size and structure.
  Total red blood count (RBC), Haemoglobin (HGB). Haematocrit (HCT), Mean Cell Volume (MCV), Mean Cell Haemoglobin (MCH), Mean Cell Haemoglobin Concentration (MCHC), and platelets (mm3).
Change Leucogram Parameters Baseline after 4, 12 and 24 weeks of intervention. | Baseline and 4, 12 and 24 weeks.
  Anticoagulated blood will be used to do the complete blood count performed using basic laboratory equipment or an automated hematology analyzer, which counts cells and collects information on their size and structure.
  Assessment of leukocyte numbers: Total WBC count (all cell types), relative (%) and absolute (cells/uL) differential leukocyte count (WBC separated by type). Neutrophils, Lymphocytes, Monocytes, Eosinophils, Basophils.
Change Circadian Rhythms Over time of Intervention. | Baseline and 4, 12 and 24 weeks.
  The first version of the Portuguese language questionnaire, "Morningness-Eveningness-Stability Scale - improved by Horne e Ostberg" (QMV-H&O), had 20 items (19 items translated from English language questionnaire and a 20th added by us).
  The total of the items is divided in three subscales, each one composed of five items: Morning Affect, Eveningness, and Distinctness. The items related to the Morning Affect subscale measure morningness preferences (early schedules), whereas the items of the Eveningness subscale assess evening preferences (late schedules). The remaining five items constitute the Distinctness subscale, that is, the amplitude dimension of this instrument. Each item is responded using a 5-points Likert scale and scored with 1-5 points, although some of them are reverse coded. The previous validation studies mentioned in the Introduction have revealed good indexes, such as Cronbach' alpha values for the three subscales ranging between 0.69 to 0.87.
Change Quality of Life Assessments Over time of Intervention. | Baseline and 4, 12 and 24 weeks.
  One of the instruments that is regularly used to measure QOL, is the World Health Organization Quality of Life instrument - 100 items (WHOQOL-100; WHOQOL Group, 1998b), a cross-culturally developed generic instrument. It was created by the World Health Organization Quality of Life Group (WHOQOL Group), that defined QOL as "an individual's perception of his/her position in life in the context of the culture and value systems in which he/she lives and in relation to his/her goals, expectations, standards and concerns" (WHOQOL group, 1995). The WHOQOL-BREF contains 26 items; one item from each of the 24 facets contained in the original WHOQOL-100 and two items were retrieved from the 'Overall QOL and General health' facet. The WHOQOL-BREF covers four domains: Physical health, Psychological health, Social relationships, and Environment.
Change Sleep Patterns Over time of Intervention. | Baseline and 4, 12 and 24 weeks.
  Sleep patterns will be evaluated using the Brazilian Portuguese Version of the Mini-Sleep Questionnaire (MSQ-BR).
  It is composed of a ten-item self-report scale that measures frequencies of sleep difficulty. Insomnia is evaluated by four questions which assess difficulty in falling asleep, mid-sleep awakenings, early awakening in the morning, and hypnotic medication use (MSQ-BR insomnia). For evaluation of hypersomnia, the questions include snoring, feeling tired upon awakening, excessive daytime sleepiness, and restless sleep (MSQ-BR hypersomnia). Answers are given on a seven-point scale ranging from 1 (never) to 7 (always). The total sum of scores is divided into four levels of sleep difficulties: 10-24 points, good sleep quality; 25-27 points, mild sleep difficulties; 28-30 points, moderate sleep difficulties; and ≥31 points, severe sleep difficulties. The total score offers an estimate of sleep quality, with higher scores reflecting more sleeping problems.
Change Sleep Quality Over Time of Intervention. | Baseline and 4, 12 and 24 weeks.
  The Pittsburgh Sleep Quality Index (PSQI) assesses sleep quality over a 1-month period. The questionnaire consists of 19 self-rated questions and 5 questions that should be answered by bedmates or roommates. The latter questions are used only for clinical information. The 19 questions categorized into 7 components, graded on a score that ranges from 0 to 3. The PSQI components are as follows: subjective sleep quality (C1), sleep latency (C2), sleep duration (C3), habitual sleep efficiency (C4), sleep disturbances (C5), use of sleeping medication(C6), and daytime dysfunction (C7). The sum of scores for these 7components yields one global score, which ranges from 0 to 21, where the highest score indicates the worst sleep quality. A global PSQIscore greater than 5 indicates major difficulties in at least 2 components or moderate difficulties in more than 3 components.
Change Sleepiness Patterns Over time of Intervention. | Baseline and 4, 12 and 24 weeks.
  Excessive daytime sleepiness (EDS) is defined as an increased propensity to fall asleep under circumstances that the affected individual and others would consider inappropriate. A Portuguese-language version of the Epworth sleepiness scale (ESS) will be applied to volunteers.
  The ESS is based on questions referring to eight such situations, some known to be very soporific; others less so. The questionnaire, which is self-administered. Subjects are asked to rate on a scale of 0-3 how likely they would be to doze off or fall asleep in the eight situations, based on their usual way of life in recent times. A distinction is made between dozing off and simply feeling tired. If a subject has not been in some of the situations recently, he is asked, nonetheless, to estimate how each might affect him.

SECONDARY OUTCOMES:
Change Body Mass Index (BMI) Over time of Intervention. | Baseline and 4, 12 and 24 weeks.
  Body Mass Index (BMI) - weight in kilograms divided by the square of height in meters (kg/m^2) .

CONTACTS AND LOCATIONS:
Overall Officials: Ana Flavia M Pessoa, Ph.D, Principal Investigator — University of São Paulo - Medical School - FMUSP
Locations (1):
- USP Medical School, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hatting M, Tavares CDJ, Sharabi K, Rines AK, Puigserver P. Insulin regulation of gluconeogenesis. Ann N Y Acad Sci. 2018 Jan;1411(1):21-35. doi: 10.1111/nyas.13435. Epub 2017 Sep 3. PMID 28868790
- [Background] Burgos-Moron E, Abad-Jimenez Z, Maranon AM, Iannantuoni F, Escribano-Lopez I, Lopez-Domenech S, Salom C, Jover A, Mora V, Roldan I, Sola E, Rocha M, Victor VM. Relationship Between Oxidative Stress, ER Stress, and Inflammation in Type 2 Diabetes: The Battle Continues. J Clin Med. 2019 Sep 4;8(9):1385. doi: 10.3390/jcm8091385. PMID 31487953
- [Background] Kutlu O, Kaleli HN, Ozer E. Molecular Pathogenesis of Nonalcoholic Steatohepatitis- (NASH-) Related Hepatocellular Carcinoma. Can J Gastroenterol Hepatol. 2018 Aug 29;2018:8543763. doi: 10.1155/2018/8543763. eCollection 2018. PMID 30228976
- [Background] Lamers F, Vogelzangs N, Merikangas KR, de Jonge P, Beekman AT, Penninx BW. Evidence for a differential role of HPA-axis function, inflammation and metabolic syndrome in melancholic versus atypical depression. Mol Psychiatry. 2013 Jun;18(6):692-9. doi: 10.1038/mp.2012.144. Epub 2012 Oct 23. PMID 23089630
- [Background] Hao H, Zheng X, Wang G. Insights into drug discovery from natural medicines using reverse pharmacokinetics. Trends Pharmacol Sci. 2014 Apr;35(4):168-77. doi: 10.1016/j.tips.2014.02.001. Epub 2014 Feb 28. PMID 24582872
- [Background] Juarez-Hernandez E, Chavez-Tapia NC, Uribe M, Barbero-Becerra VJ. Role of bioactive fatty acids in nonalcoholic fatty liver disease. Nutr J. 2016 Aug 2;15(1):72. doi: 10.1186/s12937-016-0191-8. PMID 27485440
- [Background] Sabater-Molina M, Larque E, Torrella F, Zamora S. Dietary fructooligosaccharides and potential benefits on health. J Physiol Biochem. 2009 Sep;65(3):315-28. doi: 10.1007/BF03180584. PMID 20119826
- [Background] Torres DPM, Goncalves MDPF, Teixeira JA, Rodrigues LR. Galacto-Oligosaccharides: Production, Properties, Applications, and Significance as Prebiotics. Compr Rev Food Sci Food Saf. 2010 Sep;9(5):438-454. doi: 10.1111/j.1541-4337.2010.00119.x. PMID 33467830
- [Background] Abenavoli L, Izzo AA, Milic N, Cicala C, Santini A, Capasso R. Milk thistle (Silybum marianum): A concise overview on its chemistry, pharmacological, and nutraceutical uses in liver diseases. Phytother Res. 2018 Nov;32(11):2202-2213. doi: 10.1002/ptr.6171. Epub 2018 Aug 6. PMID 30080294
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Bertolazi AN, Fagondes SC, Hoff LS, Dartora EG, Miozzo IC, de Barba ME, Barreto SS. Validation of the Brazilian Portuguese version of the Pittsburgh Sleep Quality Index. Sleep Med. 2011 Jan;12(1):70-5. doi: 10.1016/j.sleep.2010.04.020. Epub 2010 Dec 9. PMID 21145786
- [Background] Vagos P, Rodrigues PFS, Pandeirada JNS, Kasaeian A, Weidenauer C, Silva CF, Randler C. Factorial Structure of the Morningness-Eveningness-Stability-Scale (MESSi) and Sex and Age Invariance. Front Psychol. 2019 Jan 17;10:3. doi: 10.3389/fpsyg.2019.00003. eCollection 2019. PMID 30705648
- [Background] Falavigna A, de Souza Bezerra ML, Teles AR, Kleber FD, Velho MC, da Silva RC, Mazzochin T, Santin JT, Mosena G, de Braga GL, Petry FL, de Lessa Medina MF. Consistency and reliability of the Brazilian Portuguese version of the Mini-Sleep Questionnaire in undergraduate students. Sleep Breath. 2011 Sep;15(3):351-5. doi: 10.1007/s11325-010-0392-x. Epub 2010 Jul 24. PMID 20652835
- [Background] Fleck MP, Louzada S, Xavier M, Chachamovich E, Vieira G, Santos L, Pinzon V. [Application of the Portuguese version of the instrument for the assessment of quality of life of the World Health Organization (WHOQOL-100)]. Rev Saude Publica. 1999 Apr;33(2):198-205. doi: 10.1590/s0034-89101999000200012. Portuguese. PMID 10413938
- [Background] Bech P. Quality of life measurement in the medical setting. Eur Psychiatry. 1995;10 Suppl 3:83s-5s. doi: 10.1016/0924-9338(96)80085-X. PMID 19698400
- [Background] Aloe F, Pedroso A, Tavares SM. Epworth Sleepiness Scale outcome in 616 Brazilian medical students. Arq Neuropsiquiatr. 1997 Jun;55(2):220-6. doi: 10.1590/s0004-282x1997000200009. PMID 9629381
- [Background] Asnani MR, Lipps GE, Reid ME. Utility of WHOQOL-BREF in measuring quality of life in sickle cell disease. Health Qual Life Outcomes. 2009 Aug 10;7:75. doi: 10.1186/1477-7525-7-75. PMID 19664266
- [Background] Johns MW. A new method for measuring daytime sleepiness: the Epworth sleepiness scale. Sleep. 1991 Dec;14(6):540-5. doi: 10.1093/sleep/14.6.540. PMID 1798888
- [Derived] Santamarina AB, Nehmi Filho V, Freitas JA, Silva BFRBD, Gusmao AF, Olivieri EHR, Souza E, Silva SLD, Miranda DA, Demarque DP, Oliveira EDS, Otoch JP, Pessoa AFM. Nutraceutical composition (yeast beta-glucan, prebiotics, minerals, and silymarin) predicts improvement of sleep quality and metabolic parameters: A randomized pilot study. Clin Nutr ESPEN. 2024 Oct;63:476-490. doi: 10.1016/j.clnesp.2024.06.033. Epub 2024 Jul 2. PMID 39012843
- [Derived] Santamarina AB, de Freitas JA, Franco LAM, Nehmi-Filho V, Fonseca JV, Martins RC, Turri JA, da Silva BFRB, Fugi BEI, da Fonseca SS, Gusmao AF, Olivieri EHR, de Souza E, Costa S, Sabino EC, Otoch JP, Pessoa AFM. Nutraceutical blends predict enhanced health via microbiota reshaping improving cytokines and life quality: a Brazilian double-blind randomized trial. Sci Rep. 2024 May 15;14(1):11127. doi: 10.1038/s41598-024-61909-3. PMID 38750102
- [Derived] Nehmi-Filho V, Santamarina AB, de Freitas JA, Trarbach EB, de Oliveira DR, Palace-Berl F, de Souza E, de Miranda DA, Escamilla-Garcia A, Otoch JP, Pessoa AFM. Novel nutraceutical supplements with yeast beta-glucan, prebiotics, minerals, and Silybum marianum (silymarin) ameliorate obesity-related metabolic and clinical parameters: A double-blind randomized trial. Front Endocrinol (Lausanne). 2023 Jan 27;13:1089938. doi: 10.3389/fendo.2022.1089938. eCollection 2022. PMID 36778595